CLINICAL TRIAL: NCT00668720
Title: Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment in Patients With Chronic Tinnitus
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: dr. G.A. van Zanten, Department of Otorhinolaryngology, University Medical Center Utrecht
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS_tinnitus_Utrecht
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Tinnitus
Keywords: tinnitus; transcranial magnetic stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: transcranial magnetic stimulation (Magstim rapid2)
- 2 (Sham Comparator)
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation (Magstim rapid2) — Neuronavigated rTMS will be applied bilaterally to the auditory cortices, which will be identified through a structural MRI scan. Stimulation will be performed with 1 Hz frequency and an intensity of 110% motor threshold for 2000 stimuli (32 minutes) on each side, on five subsequent days.
  Other Names: Magstim rapid2
  Arms: 1
Device: sham stimulation — The official sham stimulator for the magstim rapid2 will be used. Sham stimulation will follow the same placement protocol and will also last 2x32 minutes on five subsequent days
  Arms: 2

SUMMARY:
Tinnitus is a phantom auditory perception of meaningless sound, meaning that there is registration of sound in the absence of an external or internal acoustic stimulus. It is a common problem (prevalence 7-19%) which may interfere with the ability to lead a normal life. Unfortunately, it is a very difficult symptom to treat because there are hardly any therapeutic options for the cause of tinnitus. Most therapies focus on alleviating the condition rather than treating the cause. Tinnitus is thought to be generated in the brain, as a result of functional reorganization of auditory neural pathways and tonotopic maps in the central auditory system, following damage to the peripheral auditory system. Repetitive Transcranial magnetic stimulation (rTMS) is a therapy, based on this concept of reorganization in the auditory cortex. It uses a pulsed magnetic field to disrupt the neural circuit and to thereby (temporarily) excite or inhibit certain brain areas, leading to the suppression of tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, non fluctuating, tinnitus, demonstrated by means of the diagnostic Protocol Tinnitus UMCU, of at least two months duration.
* Age ≥18 years
* Dutch speaking

Exclusion Criteria:

* Treatable cause of the tinnitus
* Use of anticonvulsant medication or other psychotherapeutic drugs
* History of epilepsy or family members with epilepsy
* Presence of active migraine
* Presence of psychiatric, severe internal or heart diseases or other neurologic diseases besides epilepsy
* Metal objects in and around body that can not be removed
* Pregnancy (will be tested on the first day of rTMS using a urine pregnancy test)
* Alcohol or drug abuse
* Prior treatment with TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Tinnitus severity with the Tinnitus Questionnaire | after treatment, 1 week, 1, 3 and 6 months

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory | after treatment, 1 week, 1, 3 and 6 months
Beck Depression Inventory | after treatment, 1 week, 1, 3 and 6 months
State Trait Anxiety Index | after treatment, 1 week, 1, 3 and 6 months
Visual Analog Scales on burden, loudness, pitch, presence, and variability of tinnitus and specific problems. | for the first three months daily and for the second three months monthly
Audiometry and tinnitus analysis (character match, pitch match, loudness match, minimal masking level, residual inhibition) | 1 week after treatment and after 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bert A van Zanten, AuD, Principal Investigator — Dept. of Otorhinolaryngology, University Medical Center Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Hoekstra CE, Versnel H, Neggers SF, Niesten ME, van Zanten GA. Bilateral low-frequency repetitive transcranial magnetic stimulation of the auditory cortex in tinnitus patients is not effective: a randomised controlled trial. Audiol Neurootol. 2013;18(6):362-73. doi: 10.1159/000354977. Epub 2013 Oct 19. PMID 24157459